CLINICAL TRIAL: NCT01106534
Title: XIENCE V® Everolimus Eluting Coronary Stent System USA Post- Approval Study (XIENCE V® USA DAPT Cohort) (XVU-AV DAPT)
Brief Title: XIENCE V® USA Dual Antiplatelet Therapy (DAPT) Cohort
Acronym: XVU-AV DAPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Baim Institute for Clinical Research (Other); Bristol-Myers Squibb (Industry); Eli Lilly and Company (Industry); Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-374C
Record Dates: First submitted 2010-04-16; First posted 2010-04-20 (Estimated); Results first posted 2016-06-28 (Estimated); Last update posted 2023-11-14 (Actual); Status verified 2023-10

CONDITIONS: Chronic Total Occlusion of Coronary Artery; Vascular Disease; Myocardial Ischemia; Coronary Artery Stenosis; Coronary Disease; Coronary Artery Disease; Coronary Restenosis
Keywords: drug eluting stents; Stents; Angioplasty; Stent thrombosis; antiplatelet treatment
MeSH Terms: conditions — Vascular Diseases; Myocardial Ischemia; Coronary Stenosis; Coronary Disease; Coronary Artery Disease; Coronary Restenosis | interventions — Aspirin; Clopidogrel; Prasugrel Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 12 month DAPT arm (Placebo Comparator): placebo + aspirin
  Interventions: Drug: placebo + aspirin; Device: XIENCE V Everolimus Eluting Coronary Stent System (XIENCE V EECSS)
- 30 month DAPT arm (Active Comparator): clopidogrel + aspirin OR prasugrel + aspirin
  Interventions: Drug: clopidogrel + aspirin OR prasugrel + aspirin; Device: XIENCE V Everolimus Eluting Coronary Stent System (XIENCE V EECSS)

INTERVENTIONS:
Drug: placebo + aspirin — This population consists of subjects enrolled in the study who are free from death, MI, stroke, repeat coronary revascularization, major bleeding, and ST 12 months after stent implantation and who are compliant with 12 months of dual antiplatelet therapy following stent implantation and who are subsequently randomized to receive 18 months of placebo treatment in addition to aspirin.
  Arms: 12 month DAPT arm
Drug: clopidogrel + aspirin OR prasugrel + aspirin — This population consists of subjects enrolled in the study who are free from death, MI, stroke, repeat coronary revascularization, major bleeding, and ST 12 months after stent implantation and who are compliant with 12 months of dual antiplatelet therapy following stent implantation and who are subsequently randomized to receive an additional 18 months of thienopyridine (clopidogrel or prasugrel) treatment in addition to aspirin.
  Other Names: Dual Antiplatelet Therapy
  Arms: 30 month DAPT arm
Device: XIENCE V Everolimus Eluting Coronary Stent System (XIENCE V EECSS) — XIENCE V Everolimus Eluting Coronary Stent System assigned to both the arms.

SUMMARY:
XIENCE V USA is a prospective, multi-center, multi-cohort postapproval study. The objectives of this study are

* To evaluate XIENCE V EECSS continued safety and effectiveness during commercial use in real world settings, and
* To support the Food and Drug Administration (FDA) dual antiplatelet therapy (DAPT) initiative. This initiative is designed to evaluate the composite of all death, myocardial infarction (MI) and stroke (MACCE) and the survival of patients that are free from Academic Research Consortium (ARC) definite or probable stent thrombosis (ST) and that have been treated with drug eluting stents (DES) and extended dual antiplatelet therapy.

DETAILED DESCRIPTION:
This prospective, multi-center, randomized, double-blind AV-DAPT study cohort is designed to collect data to support the FDA DAPT initiative. The protocol for AV-DAPT cohort is designed according to the HCRI-DAPT (NCT00977938) study protocol, Study IDE # G080186.

A total 8040 patients (5034 in initial enrollment phase and additional ~3000 patients in the second enrollment phase) enrolled in the XIENCE V USA (NCT00676520) had completed Phase I and were evaluated at 1 year.

These patients were transferred to the following cohorts in Phase II and followed-up for 1-5 years:

The long-term follow-up cohort of phase II (NCT01120379) consisted of 5020 patients from the first enrollment phase who were not transferred to the HCRI- DAPT study and remained in the study beyond 1 year.

Patients from the additional 3000 treated with the XIENCE V EECSS who are free from events (death, MI, repeat coronary revascularization, stroke, ST, or major bleeding - "severe" or "moderate" by GUSTO classification) in the first year after the index procedure, and are compliant with DAPT will be identified as prospective patients for the AV-DAPT cohort. A total of 870 Patients who are considered as part of the AV-DAPT cohort will continue with Aspirin therapy and will be randomized at 12 months post index procedure to 18 months of either active treatment with thienopyridines or placebo. Clinical follow-up will occur at 15, 24, 30 and 33 months. These patients will be followed by Abbott Vascular.

The remaining patients from the additional 3000 patients who did not participate in AV-DAPT cohort will be followed for the first year only. A study completion form will be filled out and the patients will not be followed beyond their 1 year visit.

The participants enrolled in this study will be followed by Abbott Vascular but their data will not be independently analyzed; they will only be analyzed as part of the DAPT study (NCT00977938) which is sufficiently powered for the study outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are enrolled into the XIENCE V USA Study Phase I
* The patient agrees to participate in this study by signing the Institutional Review Board (IRB) approved informed consent form. Alternatively, the patient's legally authorized representative agrees to the patient's participation in this study and signs the informed consent form.

Exclusion Criteria:

* The inability to obtain an informed consent is an exclusion criterion.

Patients must meet the following criteria to be eligible for randomization in the study:

* Patient is "12 Month Clear": "12-Month Clear" patients are free from death, MI, stroke, repeat coronary revascularization, major bleeding - "severe" or "moderate" by GUSTO classification, and ST 12 months after stent implantation. Staged PCI is allowed (same stent type as index); repeat PCI and peri-procedural myocardial infarction occurring with the index procedure or repeat procedure within the first 6 weeks will not be considered exclusionary events for the definition of "12 Month Clear".
* Patient is "DAPT Compliant": During the open label portion of this study (time 0-12 months), a patient is considered compliant with the thienopyridine therapy for the purposes of eligibility if they take between 80% and 120% of the prescribed drug in a given period without an interruption of therapy longer than 14 days. This information will be ascertained via data collected at the patient interviews at 6 and 12 months post-procedure. Compliance at both time points is required to be considered "clear".
* Patient completes 1 year visit within ± 30 days window.

Patients will be excluded from randomization if any of the following criteria are met:

* Pregnant women.
* Switched thienopyridine type or dose within 6 months prior to randomization. Note: Thienopyridine switching during the open label portion of this study is discouraged.
* PCI or cardiac surgery between 6 weeks post index procedure and randomization.
* Planned surgery necessitating discontinuation of antiplatelet therapy within the 21 months following randomization.
* Current medical condition with a life expectancy of less than 3 years.
* Patients on warfarin or similar anticoagulant therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 870 (Actual)
Dates: Start 2009-08; Primary Completion 2015-02 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Hermiller, MD, Principal Investigator — Heart Center of Indianapolis; Mitch Krucoff, MD, Principal Investigator — Duke University
Locations (144):
- United States (144):
  - Birmingham Heart Clinic, PC, Birmingham, Alabama
  - Thomas Hospital, Fairhope, Alabama
  - Scottsdale Healthcare, Scottsdale, Arizona
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - California Cardiovascular Consultants, Fremont, California
  - FACT/ Los Angeles Cardiology, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - Eisenhower Medical Center, Desert Cardiology Center, Rancho Mirage, California
  - Regional Cardiology Associates, Sacramento, California
  - Salinas Valley Memorial Healthcare System, Salinas, California
  - Sansum Clinic, Santa Barbara, California
  - Torrance Memorial Medical Center, Torrance, California
  - The Medical Center of Aurora, Aurora, Colorado
  - St. Anthony's Central Hospital, Denver, Colorado
  - St. Vincent's Medical Center, Norwalk, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Brandon Regional Hospital, Brandon, Florida
  - Morton Plant Hospital, Clearwater, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Cardiology Partners Clinical Research Institute (Formerly Palm Beach Gardens Medical Center), Wellington, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - University Hospital Augusta Cardiology Clinic, Augusta, Georgia
  - NE Georgia Medical Center, Gainesville, Georgia
  - WellStar Kennestone Hospital, Marietta, Georgia
  - Midwest Heart Foundation, Lombard, Illinois
  - Heart Care Midwest (OSF/St Francis), Peoria, Illinois
  - St. John's Hospital / Prairie Education & Research Cooperative, Springfield, Illinois
  - Elkhart Midwest Cardiovascular Research & Education Foundation, Elkhart, Indiana
  - The Care Group at Methodist, Indianapolis, Indiana
  - St. Francis Hospital and Health Centers, Indianapolis, Indiana
  - Indiana Heart Hospital, Indianapolis, Indiana
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - Galichia Heart Hospital, Wichita, Kansas
  - Central Baptist Hospital, Lexington, Kentucky
  - Northeast Cardiology Associates, Bangor, Maine
  - Maine Cardiology Associates, South Portland, Maine
  - Union Memorial Hospital, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Washington Adventist Hospital, Takoma Park, Maryland
  - St. Joseph Medical Center, Towson, Maryland
  - Boston Medical Center East, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - St John Hospital & Medical Center, Detroit, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - St. Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Michigan Cardio Vascular Institute at St. Mary's of MI, Saginaw, Michigan
  - Covenant Medical Center, INC., Saginaw, Michigan
  - Lakeland Hospital St. Joseph, Saint Joseph, Michigan
  - St. Joseph Mercy Hospital, Ypsilanti, Michigan
  - North Memorial Medical Center, Minneapolis, Minnesota
  - Mercy Hospital, Minneapolis, Minnesota
  - St. Paul Heart Clinic, Saint Paul, Minnesota
  - Southern Heart Center, Hattiesburg, Mississippi
  - Jackson Heart Clinic, Jackson, Mississippi
  - St. Luke's Hospital, Kansas City, Missouri
  - North Kansas City Hospital, North Kansas City, Missouri
  - St. John's Research Institute, Inc., St. John's Hospital, Springfield, Missouri
  - Barnes Jewish Hospital, St Louis, Missouri
  - Billings Clinic Research Center, Billings, Montana
  - Dartmouth Hitchock Medical Center, Lebanon, New Hampshire
  - Englewood Hospital & Medical Center, Englewood, New Jersey
  - Hackensack Medical Center, Hackensack, New Jersey
  - CADV, Haddon Heights, New Jersey
  - St. Joseph's Regional Medical Center, Paterson, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - St. Peters Hospital, Albany, New York
  - Buffalo Heart group, Buffalo, New York
  - Mount Sinai Medical Center, New York, New York
  - Rochester Cardiopulmonary Group, Rochester, New York
  - Stony Brook Hospital and Medical Center, Stony Brook, New York
  - St. Joseph's Hospital Health Center, Syracuse, New York
  - Jack D. Weiler Hospital of Montefiore Medical Center, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Mid Carolina Cardiology, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Gaston Memorial Hospital, Gastonia, North Carolina
  - High Point Regional Health System, High Point, North Carolina
  - WakeMed Hospital, Raleigh, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Altru Health System, Grand Forks, North Dakota
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - North Ohio Research LTD, Elyria Regional Medical Center, Elyria, Ohio
  - Fairview Hospital, Fairview Park, Ohio
  - The Toledo Hospital-Jobst Vascular Center, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Cardiology Associates of Southeastern Ohio, Inc, Zanesville, Ohio
  - Midwest Regional Medical Center, Midwest City, Oklahoma
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Integris Baptist Medical, Inc., Oklahoma City, Oklahoma
  - Hillcrest Medical Center, Tulsa, Oklahoma
  - Sacred Heart Medical Center, Eugene, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Tri-State Medical Group, Beaver, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Franklin County Heart Center at Summit Cardiology, Chambersburg, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Harrisburg Hospital / Pinnacle Health, Harrisburg, Pennsylvania
  - Lancaster Heart & Stroke Foundation, Lancaster, Pennsylvania
  - Hahnemann Hospital, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - The Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Holy Spirit Hospital, Wormleysburg, Pennsylvania
  - Main Line Health Heart Center/The Lankenau Hospital, Wynnewood, Pennsylvania
  - York Hospital, York, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - AnMed Health, Anderson, South Carolina
  - Providence Hospital-SC, Columbia, South Carolina
  - Sanford USD Medical Center, Sioux Falls, South Dakota
  - Memorial Health System, Chattanooga, Tennessee
  - West Clinic d/b/a Memphis Heart Clinic, Memphis, Tennessee
  - Centennial Heart Cardiovascular Consultants, LLC., Nashville, Tennessee
  - St. Thomas Hospital, Nashville, Tennessee
  - Vanderbilt Vniversity Medical Center, Nashville, Tennessee
  - Amarillo Heart Clinical Research Institute, Amarillo, Texas
  - Capital Cadiovascular Specialists, Austin, Texas
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - The Methodist Hospital, Houston, Texas
  - Lubbock Heart Hospital, Lubbock, Texas
  - Permian Research Foundation, Odessa, Texas
  - South Texas Methodist Hospital, San Antonio, Texas
  - Intermountain Medical Center, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Virginia Cardiovascular Consultants, Fredericksburg, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Carilion Roanoke Memorial, Roanoke, Virginia
  - Overlake Hospital Medical Center, Bellevue, Washington
  - Providence Everett Medical Center, Everett, Washington
  - St. Joseph's Tacoma, Tacoma, Washington
  - St Mary's Medical Hospital, Huntington, West Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Wisconsin Heart Hospital, Wauwatosa, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Additional 3000 patients were enrolled in the second enrollment phase and had completed phase I at 1 year. In phase II, 870 patients from these were transferred to AV-DAPT cohort and followed from 1 year to 33 months, and the remaining who did not participate in AV-DAPT cohort will be followed for the first year only.
Pre-assignment Details: Outcome measures of participants of XIENCE V USA trial of phase I followed up until 1 year from index procedure are available in the study with ID NCT00676520.
  Outcome measures of participants belonging to XIENCE V USA long-term follow-up cohort of phase II (followed up from year 1 to year 5) are available in the study with ID NCT01120379.
Groups:
- Second Enrollment Phase of XIENCE V® USA: Additional 3000 patients recruited in the second enrollment phase treated with the XIENCE V EECSS who are free from events (death, MI, repeat coronary revascularization, stroke, ST, or major bleeding - "severe" or "moderate" by GUSTO classification) in the first year after the index procedure, and are compliant with DAPT will be identified as prospective patients for the AV-DAPT cohort. A total of 870 Patients who are considered as part of the AV-DAPT cohort will continue with Aspirin therapy and will be randomized at 12 months post index procedure to 18 months of either active treatment with thienopyridines or placebo. Clinical follow-up will occur at 15, 24, 30 and 33 months. These patients will be followed by Abbott Vascular.
Period: Overall Study
Arm/Group | Second Enrollment Phase of XIENCE V® USA
Started | 2997
Completed | 2960
Not Completed | 37
Not completed — Withdrawal by Subject | 18
Not completed — Lost to Follow-up | 2
Not completed — Death | 16
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are provided for 2997 patients recruited in the second enrollment phase.
Arm/Group | Second Enrollment Phase of XIENCE V® USA
Number analyzed (Participants) | 2997
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.27 (10.39)
Age, Customized [Number; unit: participants]
  < 65 years | 1587
  >= 65 to < 75 years | 922
  >= 75 years | 488
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 870
  Male | 2127
Race/Ethnicity, Customized [Number; unit: participants] — Patient may be counted in more than one category
  participants
    American Indian or Alaskan Native | 23
    Asian | 49
    Black or African Heritage | 231
    Native Hawaiian or Pacific Islander | 7
    White | 2577
    Hispanic or Latino | 117
    Other | 15

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Composite of All Death, MI and Stroke (Defined as MACE)
Time Frame: 12-33 months post-stent
Population: Participants enrolled in the study will be followed by Abbott Vascular but their data will not be independently analyzed; they will only be analyzed as part of the DAPT study (NCT00977938) which is sufficiently powered for the study outcomes.
Arm/Group | 12 Month DAPT Arm | 30 Month DAPT Arm
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Incidence of ARC Definite or Probable ST
Time Frame: 12-33 months post-stent
Population: as for outcome 1
Arm/Group | 12 Month DAPT Arm | 30 Month DAPT Arm
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Major Bleeding (GUSTO Classification, Severe and Moderate Bleeding Combined)
Time Frame: 12-33 months post-stent
Population: as for outcome 1
Arm/Group | 12 Month DAPT Arm | 30 Month DAPT Arm
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: MACE for ITT Population
Time Frame: 12 through 30 months
Population: as for outcome 1
Arm/Group | 12 Month DAPT Arm | 30 Month DAPT Arm
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: ST for ITT Population
Time Frame: 12 through 30 months
Population: as for outcome 1
Arm/Group | 12 Month DAPT Arm | 30 Month DAPT Arm
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Major Bleeding for ITT Population
Time Frame: 12 through 30 months
Population: as for outcome 1
Arm/Group | 12 Month DAPT Arm | 30 Month DAPT Arm
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: MACE for Treatment Population
Time Frame: 12 through 30 months and 12 through 33 months
Population: as for outcome 1
Arm/Group | 12 Month DAPT Arm | 30 Month DAPT Arm
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: ST for Treatment Population
Time Frame: 12 through 30 months and 12 through 33 months
Population: as for outcome 1
Arm/Group | 12 Month DAPT Arm | 30 Month DAPT Arm
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Major Bleeding for Treatment Population
Time Frame: 12 through 30 months and 12 through 33 months
Population: as for outcome 1
Arm/Group | 12 Month DAPT Arm | 30 Month DAPT Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 5 years
Description: Adverse events were not be reported here as the participants enrolled in this study will be followed by Abbott Vascular but their data will not be independently analyzed; they will only be analyzed as part of the DAPT study (NCT00977938) which is sufficiently powered for the study outcomes.
Groups:
- Second Enrollment Phase of XIENCE V® USA: The participants enrolled in this study will be followed by Abbott Vascular but their data will not be independently analyzed; they will only be analyzed as part of the DAPT study (NCT00977938) which is sufficiently powered for the study outcomes.
Arm/Group | Second Enrollment Phase of XIENCE V® USA
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The participants enrolled in this study will be followed by Abbott Vacular but their data will not be independently analyzed; they will only be analyzed as part of the DAPT study (NCT00977938) which is sufficiently powered for the outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days